CLINICAL TRIAL: NCT03777436
Title: A Phase 3, Multicenter, Randomized, Placebo-Controlled, Double Blind-Study of the Efficacy and Safety of Apremilast (CC-10004) in Subjects With Moderate to Severe Genital Psoriasis
Brief Title: An Efficacy and Safety Study of Apremilast (CC-10004) in Subjects With Moderate to Severe Genital Psoriasis
Acronym: DISCREET
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CC-10004-PSOR-025; U1111-1224-6850 (Registry Identifier: WHO); 2018-002608-15 (EudraCT Number)
Expanded Access: NCT03740516 (No longer available)
Record Dates: First submitted 2018-12-14; First posted 2018-12-17 (Actual); Results first posted 2022-12-15 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Psoriasis
Keywords: Genital Psoriasis; CC-10004; Apremilast; Plaque Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — apremilast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A- Apremilast with Placebo (Experimental): Subjects randomized to the apremilast 30 mg BID treatment group will receive apremilast 30 mg tablets orally twice daily for the first 16 weeks Subjects randomized to the placebo treatment group will receive placebo tablets (identical in appearance to apremilast 30 mg tablets) orally twice daily for the first 16 weeks
  Interventions: Drug: Apremilast; Other: Placebo
- Arm B - Apremilast 30 mg (Experimental): All subjects will receive apremilast 30 mg tablets orally twice daily after the Week 16 Visit through the end of the Apremilast Extension Phase of the study
  Interventions: Drug: Apremilast

INTERVENTIONS:
Drug: Apremilast — Oral
  Other Names: CC-10004, Otezla
Other: Placebo — Oral
  Arms: Arm A- Apremilast with Placebo

SUMMARY:
This Phase 3 multicenter, randomized, placebo-controlled, double-blind study is designed to evaluate the efficacy and safety of apremilast in subjects with moderate to severe genital psoriasis (modified sPGA-G ≥3, moderate or severe).

Approximately 286 subjects with moderate to severe genital psoriasis will be randomized 1:1 to receive either apremilast 30 mg BID or placebo for the first 16 weeks.

DETAILED DESCRIPTION:
The study will consist of four phases:

* Screening Phase - up to 35 days
* Double-blind Placebo-controlled Phase - Weeks 0 to 16

  - Subjects will be randomly assigned to either apremilast 30 mg tablets orally BID or placebo tablets (identical in appearance to apremilast 30 mg tablets) orally BID.
* Apremilast Extension Phase - Weeks 16 to 32

  - All subjects will be switched to (or continue with) apremilast 30 mg BID. All subjects will maintain this dosing through Week 32.
* Observational Follow-up Phase - 4 weeks - Four-week Post-Treatment Observational Follow-up Phase for all subjects who complete the study or discontinue the study early.

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy the following criteria to be enrolled in the study:

1. Subject is ≥ 18 years of age at the time of signing the informed consent form (ICF).
2. Subject must have a diagnosis of chronic plaque psoriasis for at least 6 months prior to signing the ICF.
3. Subject must have a diagnosis of moderate or severe psoriasis of the genital area at Screening and Baseline.
4. Subject must have a diagnosis of moderate or severe psoriasis at Screening and Baseline.
5. Subject must have plaque psoriasis (BSA ≥ 1%) in a non-genital area at both Screening and Baseline.
6. Subject must have been inadequately controlled with or intolerant of topical therapy, or topical therapy is inappropriate for the treatment of psoriasis affecting the genital area.
7. Subject must be in good health (except for psoriasis) as judged by the investigator, based on medical history, physical examination, clinical laboratories, and urinalysis.
8. Subject must meet laboratory criteria

Exclusion Criteria:

The presence of any of the following will exclude a subject from enrollment:

1. Subject has any significant medical condition or laboratory abnormality, that would prevent the subject from participating in the study.
2. Subject has any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study.
3. Subject has positive Hepatitis B surface antigen or anti-hepatitis C antibody at Screening.
4. Subject has active tuberculosis (TB) or a history of incompletely treated TB.
5. Subject has prior history of suicide attempt at any time in the subject's life time prior to signing the informed consent and randomization, or major psychiatric illness requiring hospitalization within the last 3 years prior to signing the informed consent.
6. Subject has current or planned therapies that may have a possible effect on psoriasis of the body and/or genital area during the course of the treatment phase of the trial
7. Subject had prior treatment with apremilast.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 289 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2021-09-23 (Actual); Study Completion 2022-02-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (52):
- United States (26):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - First OC Dermatology, Fountain Valley, California
  - Clinical Science Institute, Santa Monica, California
  - Glick Skin Institute, Margate, Florida
  - International Dermatology Research, Inc, Miami, Florida
  - Skin Care Physicians of Georgia, Macon, Georgia
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - Adult and Pediatric Dermatology, Overland Park, Kansas
  - ActivMed Practices and Research Inc, Beverly, Massachusetts
  - Brigham and Womens Hospital, Boston, Massachusetts
  - J Woodson Dermatology and Associates, Henderson, Nevada
  - Las Vegas Dermatology, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - ActivMed, Portsmouth, New Hampshire
  - Stony Brook Dermatology Associates, Stony Brook, New York
  - Dermatology Consulting Services, High Point, North Carolina
  - Oakview Dermatology, Athens, Ohio
  - Ohio State University Medical Center, Gahanna, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Paddington Testing Company Inc, Philadelphia, Pennsylvania
  - Clinical Partners LLC, Johnston, Rhode Island
  - Center for Clinical Studies, Houston, Texas
  - Austin Institute for Clinical Research, Pflugerville, Texas
  - Virginia Clinical Research Inc, Norfolk, Virginia
  - Bellevue Dermatology Clinic, Bellevue, Washington
  - Dermatology Center for Skin Health, Morgantown, West Virginia
- Belgium (3):
  - Centre Hospitalier Universitaire Saint Pierre, Brussels
  - Cliniques Universitaires St Luc, Brussels
  - UZ Leuven, Leuven
- Canada (5):
  - Guenther Dermatology Research Centre, London, Ontario
  - Lynderm Research Inc, Markham, Ontario
  - K Papp Clinical Research, Waterloo, Ontario
  - Dre Angelique Gagne-Henley M.D. Inc, Saint-Jérôme, Quebec
  - Skincare Studio, St. John's
- France (4):
  - Hopital Claude Huriez CHRU Lille, Lille
  - CHU de Nice Archet I, Nice
  - Centre Hospitalier Universitaire (CHU) de Bordeaux - Hopital Saint-Andre, Pessac
  - Larrey University Hospital, Toulouse
- Germany (6):
  - ISA - Interdisciplinary Study Association GmbH, Berlin
  - Universitaetsklinikum Bonn, Bonn
  - Hautklinik Universitatsklinikum Erlangen, Erlangen
  - Universitatsklinikum Frankfurt, Frankfurt am Main
  - Universitaetsklinikum Schleswig-Holstein, Campus Luebeck, Lübeck
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
- Italy (7):
  - Ospedali Riuniti di Ancona, Ancona
  - Presidio Ospedaliero della Misericordia, Grosseto
  - Azienda Sanitaria Locale 1 Ospedale Regionale San Salvatore, LAquila
  - Azienda Ospedaliera Di Padova, Padua
  - Azienda Ospedaliera Bianchi Melacrino Morelli, Reggio Calabria
  - Universita degli Studi di Roma La Sapienza Ospedale A Fiorini di Terracina, Terracina
  - Azienda Sanitaria Universitaria Integrata di Trieste, Trieste
- GCM Medical Group, PSC, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- [Background] Merola JF, Parish LC, Guenther L, Lynde C, Lacour JP, Staubach P, Cheng S, Paris M, Picard H, Deignan C, Jardon S, Chen M, Papp KA. Efficacy and safety of apremilast in patients with moderate-to-severe genital psoriasis: Results from DISCREET, a phase 3 randomized, double-blind, placebo-controlled trial. J Am Acad Dermatol. 2024 Mar;90(3):485-493. doi: 10.1016/j.jaad.2023.10.020. Epub 2023 Oct 16. PMID 37852306
- [Derived] Merola JF, Guenther L, Lynde C, Papp KA, Parish LC, Yamauchi P, Cheng S, Amouzadeh H, Deignan C, Jardon S, Chen M, Pinter A. Results from the 32-week, phase 3 DISCREET study of apremilast in patients with moderate to severe genital psoriasis. J Eur Acad Dermatol Venereol. 2026 Feb;40(2):274-284. doi: 10.1111/jdv.70110. Epub 2025 Dec 10. PMID 41369155
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 49 centers in Belgium, Canada, France, Germany, Italy, and the United States from February 2019 to February 2022.
Pre-assignment Details: Participants were randomized in a 1:1 ratio to receive either apremilast or matched placebo for the first 16 weeks (Placebo-controlled Phase) of the study. At Week 16, eligible participants may have continued on active treatment by entering a 16-week extension phase (Apremilast Extension Phase). Total treatment duration = 32 weeks.
Groups:
- Placebo-controlled Phase: Placebo: Participants received placebo as oral tablets twice daily (BID) for up to 16 weeks (Week 0 to Week 16).
- Placebo-controlled Phase: Apremilast 30 mg: Participants received apremilast 30 mg as oral tablets BID for up to 16 weeks (Week 0 to Week 16).
- Apremilast Extension Phase: Apremilast 30 mg: Eligible participants who completed the Placebo-controlled Phase entered the Apremilast Extension Phase and received apremilast 30 mg as oral tablets BID for up to an additional 16 weeks (Week 16 to Week 32).
Period: Placebo-controlled Phase
Arm/Group | Placebo-controlled Phase: Placebo | Placebo-controlled Phase: Apremilast 30 mg | Apremilast Extension Phase: Apremilast 30 mg
Started | 146 | 143 | 0 (This arm was not included in the Placebo-controlled Phase.)
Took at Least 1 Dose of Investigational Product (IP) | 145 | 143 | 0 (This arm was not included in the Placebo-controlled Phase.)
Completed | 111 | 119 | 0 (This arm was not included in the Placebo-controlled Phase.)
Not Completed | 35 | 24 | 0
Not completed — Adverse Event | 8 | 10 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0
Not completed — Withdrawal by Subject | 19 | 3 | 0
Not completed — Non-compliance with study drug | 0 | 2 | 0
Not completed — Lost to Follow-up | 7 | 7 | 0
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Due to COVID-19 control measures | 1 | 0 | 0
Period: Apremilast Extension Phase
Arm/Group | Placebo-controlled Phase: Placebo | Placebo-controlled Phase: Apremilast 30 mg | Apremilast Extension Phase: Apremilast 30 mg
Started | 0 (This arm was not included in the Apremilast Extension Phase.) | 0 (This arm was not included in the Apremilast Extension Phase.) | 229 (1 participant did not enter the Apremilast Extension Phase as they were lost to follow-up.)
Took at Least 1 Dose of IP | 0 (This arm was not included in the Apremilast Extension Phase.) | 0 (This arm was not included in the Apremilast Extension Phase.) | 228
Completed | 0 (This arm was not included in the Apremilast Extension Phase.) | 0 (This arm was not included in the Apremilast Extension Phase.) | 201
Not Completed | 0 | 0 | 28
Not completed — Adverse Event | 0 | 0 | 6
Not completed — Lack of Efficacy | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 13
Not completed — Lost to Follow-up | 0 | 0 | 7
Not completed — Miscellaneous | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) analysis set consisted of all participants who are randomized regardless of whether the participant received investigational product (IP).
Groups:
- Placebo-controlled Phase: Placebo: Participants received placebo as oral tablets BID for up to 16 weeks (Week 0 to Week 16).
- Total: Total of all reporting groups
Arm/Group | Placebo-controlled Phase: Placebo | Placebo-controlled Phase: Apremilast 30 mg | Total
Number analyzed (Participants) | 146 | 143 | 289
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.4 (14.38) | 43.5 (13.36) | 45.0 (13.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 43 | 87
  Male | 102 | 100 | 202
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 18 | 31
  Not Hispanic or Latino | 131 | 125 | 256
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 8 | 4 | 12
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 3 | 6 | 9
  White | 131 | 131 | 262
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 5
Modified Static Physician Global Assessment of Genitalia (sPGA-G) Score [Count of Participants; unit: Participants] — The modified sPGA-G is the assessment by the Investigator of the participant's psoriasis lesions' overall disease severity in the genital area at the time of evaluation. The modified sPGA-G is a 5-point scale ranging from clear (0), almost clear (1), mild (2), moderate (3), to severe (4), incorporating an assessment of the severity of the three primary signs of the disease: erythema, plaque elevation, and scaling.
  Participants
    3 (Moderate) | 128 | 123 | 251
    4 (Severe) | 18 | 20 | 38

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Modified sPGA-G Response at Week 16
Description: The modified sPGA-G is the assessment by the Investigator of the participant's psoriasis lesions' overall disease severity in the genital area at the time of evaluation. The modified sPGA-G is a 5-point scale ranging from clear (0), almost clear (1), mild (2), moderate (3), to severe (4), incorporating an assessment of the severity of the 3 primary signs of the disease: erythema, plaque elevation, and scaling.
  A modified sPGA-G response is defined as modified sPGA-G score of clear (0) or almost clear (1) and with ≥ 2-point reduction from Baseline at Week 16.
  Missing values were imputed using the multiple imputation (MI) method. Two-sided 95% confidence intervals (CIs) for the within-group proportions were based on the Wilson-score method.
Time Frame: Baseline and Week 16 of the Placebo-controlled Phase
Population: The ITT analysis set consisted of all participants who are randomized regardless of whether the participant received IP.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo-controlled Phase: Placebo | Placebo-controlled Phase: Apremilast 30 mg
Number analyzed (Participants) | 146 | 143
Percentage of participants | 19.5 [12.7 to 26.3] | 39.6 [31.2 to 48.0]
Statistical Analysis 1: Comparison: Placebo-controlled Phase: Placebo vs Placebo-controlled Phase: Apremilast 30 mg; Test type: Superiority; p = 0.0003, Cochran-Mantel-Haenszel; Adjusted difference = 20.1, 95% CI 2-sided [9.2 to 30.9] — Adjusted difference is the weighted average of the treatment differences across the strata with the Cochran-Mantel-Haenszel (CMH) weights. 2-sided 95% CIs based on the stratified Newcombe method. Two-sided p-values were based on the CMH test

2. Secondary Outcome: Percentage of Participants With a Static Physician Global Assessment (sPGA) Response at Week 16
Description: The sPGA is the assessment by the Investigator of the overall disease severity at the time of evaluation. The sPGA is a 5-point scale ranging from 0 (clear), 1 (almost clear), 3 (moderate) to 4 (severe), incorporating an assessment of the severity of the 3 primary signs of the disease: erythema, scaling and plaque elevation.
  An sPGA response is defined as sPGA score of clear (0) or almost clear (1) and with ≥ 2-point reduction from Baseline at Week 16.
  Missing values were imputed using the MI method. Two-sided 95% CIs for the within-group proportions were based on the Wilson-score method.
Time Frame: Baseline and Week 16 of the placebo-controlled phase
Population: The ITT analysis set consisted of all participants who are randomized regardless of whether the participant received IP.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo-controlled Phase: Placebo | Placebo-controlled Phase: Apremilast 30 mg
Number analyzed (Participants) | 146 | 143
Percentage of participants | 6.9 [2.7 to 11.2] | 22.2 [15.0 to 29.3]
Statistical Analysis 1: Comparison: Placebo-controlled Phase: Placebo vs Placebo-controlled Phase: Apremilast 30 mg; Test type: Superiority; p = 0.0004, Cochran-Mantel-Haenszel; Adjusted difference = 15.2, 95% CI 2-sided [6.9 to 23.6] — Adjusted difference is the weighted average of the treatment differences across the strata with the CMH weights. 2-sided 95% CIs based on the stratified Newcombe method. Two-sided p-values were based on the CMH test

3. Secondary Outcome: Percentage of Participants With a Genital Psoriasis Itch Numeric Rating Scale (GPI-NRS) Response at Week 16
Description: The GPI-NRS is a self-reported measure where participants were asked to assess their psoriasis symptoms in the genital area and select a number on a scale of 0-10, where 0 represents no itch, and 10 represents the worst imaginable itch.
  A GPI-NRS response is defined as ≥ 4 point reduction (improvement) from Baseline.
  Missing values were imputed using the MI method. Two-sided 95% CIs for the within-group proportions were based on the Wilson-score method.
Time Frame: Baseline and Week 16 of the placebo-controlled phase
Population: ITT analysis set with Baseline GPI-NRS score ≥ 4.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo-controlled Phase: Placebo | Placebo-controlled Phase: Apremilast 30 mg
Number analyzed (Participants) | 121 | 122
Percentage of participants | 19.6 [11.9 to 27.4] | 47.3 [37.9 to 56.6]
Statistical Analysis 1: Comparison: Placebo-controlled Phase: Placebo vs Placebo-controlled Phase: Apremilast 30 mg; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Adjusted difference = 27.4, 95% CI 2-sided [15.4 to 39.3] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Change From Baseline in Affected Body Surface Area (BSA) at Week 16
Description: The BSA is a measurement of involved skin over the whole body. The overall BSA affected by psoriasis is estimated based on the palm area of the participant's hand. The surface area of the whole body is made up of approximately 100 palms or "handprints" (each entire palmar surface or "handprint" equates to approximately 1% of total BSA).
  A negative change from Baseline indicates a reduction of affected BSA.
  Based on mixed-effect model for repeated measures (MMRM) model.
Time Frame: Baseline and Week 16 of the placebo-controlled phase
Population: ITT analysis set with Baseline and at least one post-baseline value at Week 16.
Measure: Least Squares Mean (Standard Error); unit: Change in percentage of affected BSA
Arm/Group | Placebo-controlled Phase: Placebo | Placebo-controlled Phase: Apremilast 30 mg
Number analyzed (Participants) | 111 | 120
Change in percentage of affected BSA | -0.79 (0.669) | -4.12 (0.664)
Statistical Analysis 1: Comparison: Placebo-controlled Phase: Placebo vs Placebo-controlled Phase: Apremilast 30 mg; Test type: Superiority; p = 0.0005, MMRM; Least squares mean difference = -3.33, 95% CI 2-sided [-5.18 to -1.47], Standard Error of Mean 0.942 — Based on MMRM model

5. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) at Week 16
Description: The DLQI is a 10 item questionnaire dealing with the participant's skin. With the exception of Item Number 7, the participant responds on a four-point scale, ranging from 0 (not at all) to 3 (very much). Item Number 7 is a multi-part item, the first part of which ascertains whether the participant's skin prevented them from working or studying (Yes or No), and if "No," then the participant is asked how much of a problem the skin has been at work or study over the past week, with response alternatives being 0 (not at all), 1 (a little) and 2 (a lot).
  Total scores have a possible range of 0-30, where 0 represents the best score, and 30 represents the worst health-related quality of life.
  A negative change from Baseline indicates an improvement in health-related quality of life scores.
Time Frame: Baseline and Week 16 of the placebo-controlled phase
Population: ITT analysis set with Baseline and at least one post-baseline value at Week 16.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo-controlled Phase: Placebo | Placebo-controlled Phase: Apremilast 30 mg
Number analyzed (Participants) | 107 | 117
Scores on a scale | -2.6 (0.57) | -5.3 (0.55)
Statistical Analysis 1: Comparison: Placebo-controlled Phase: Placebo vs Placebo-controlled Phase: Apremilast 30 mg; Test type: Superiority; p = 0.0008, MMRM; Least squares mean difference = -2.7, 95% CI 2-sided [-4.2 to -1.1], Standard Error of Mean 0.79 — Based on MMRM model

6. Secondary Outcome: Change From Baseline in Genital Psoriasis Symptoms Scale (GPSS) Total Score at Week 16
Description: The GPSS is a self-reported measure where participants were asked to assess each of their psoriasis symptoms (itch, pain, discomfort, stinging, burning, redness, scaling, and cracking) in the genital area and select a number on a scale of 0-10, where 0 represents no symptoms, and 10 represents the worst imaginable.
  Results from each symptom assessment were summed to generate a total GPSS score ranging from 0 (no genital psoriasis symptoms) to 80 (worst imaginable genital psoriasis symptoms).
  A negative change from Baseline indicates an improvement in genital psoriasis symptoms.
Time Frame: Baseline and Week 16 of the placebo-controlled phase
Population: ITT analysis set with Baseline and at least one post-baseline value at Week 16.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo-controlled Phase: Placebo | Placebo-controlled Phase: Apremilast 30 mg
Number analyzed (Participants) | 107 | 116
Score on a scale | -5.3 (1.85) | -20.5 (1.83)
Statistical Analysis 1: Comparison: Placebo-controlled Phase: Placebo vs Placebo-controlled Phase: Apremilast 30 mg; Test type: Superiority; p < 0.0001, MMRM; Difference = -15.1, 95% CI 2-sided [-20.3 to -10.0], Standard Error of Mean 2.60 — Based on MMRM model

ADVERSE EVENTS:
Time Frame: Up to a maximum of 41.4 weeks
Description: The safety analysis set consisted of all participants who were randomized and received at least one dose of IP.
Arm/Group | Placebo-controlled Phase: Placebo | Placebo-controlled Phase: Apremilast 30 mg | Apremilast Extension Phase: Apremilast 30 mg
All-Cause Mortality (participants affected / at risk) | 0/145 | 0/143 | 0/229
Serious Adverse Events (participants affected / at risk) | 2/145 | 3/143 | 2/229
Other Adverse Events (participants affected / at risk) | 39/145 | 73/143 | 53/229
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo-controlled Phase: Placebo (N=145) | Placebo-controlled Phase: Apremilast 30 mg (N=143) | Apremilast Extension Phase: Apremilast 30 mg (N=229)
Appendicitis (Infections and infestations) | 0 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo-controlled Phase: Placebo (N=145) | Placebo-controlled Phase: Apremilast 30 mg (N=143) | Apremilast Extension Phase: Apremilast 30 mg (N=229)
Diarrhoea (Gastrointestinal disorders) | 12 | 37 | 27
Nausea (Gastrointestinal disorders) | 11 | 32 | 17
Nasopharyngitis (Infections and infestations) | 12 | 12 | 11
Headache (Nervous system disorders) | 16 | 33 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2021-03-03): https://cdn.clinicaltrials.gov/large-docs/36/NCT03777436/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-22): https://cdn.clinicaltrials.gov/large-docs/36/NCT03777436/SAP_001.pdf